CLINICAL TRIAL: NCT00295620
Title: A Prospective, Randomized, Open, Multicentre Phase III-study to Assess the Efficacy of Secondary Adjuvant Endocrine Anastrozole Therapy for 2 Further Yrs vs 5 Further Yrs in Patients With HR +ve Breast Cancer After 5-yr Primary Adjuvant Endocrine Therapy
Brief Title: Secondary Adjuvant Long Term Study With Arimidex
Acronym: SALSA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1033AU/0003; ABCSG 16; D5392L00016; SALSA
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
Keywords: Hormone receptor positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Anastrozol (Experimental): 1 mg per day for 2 years
  Interventions: Drug: Anastrozole
- Arm B: Anastrozol (Experimental): 1 mg per day for 5 years
  Interventions: Drug: Anastrozole

INTERVENTIONS:
Drug: Anastrozole — 1mg tablet daily
  Other Names: Arimidex

SUMMARY:
The study assesses the effect of further 2 years vs further 5 years of adjuvant treatment with anastrozole after initial 5 years of adjuvant endocrine therapy.

DETAILED DESCRIPTION:
ABCSG 16 S.A.L.S.A is assessing the effect of further 2 years vs further 5 years of adjuvant treatment with anastrozole after initial 5 years of adjuvant endocrine therapy. S.A.L.S.A. is a randomized open multicentered phase III study comparing the efficacy of secondary adjuvant endokrine treatment of Arimidex® (Anastrozol) for 2 or 5 years after primary adjuvant endokrine therapy in patients with hormonreceptor positive mammakarzinom. Patients are examined at screening, after 6 months, then every year until 5 years. The subsequent yearly follow up with mammographie and clinical examination ends 10 years after the screening. S.A.L.S.A. started in February 2004 and has recruited 3484 patients until June 2010 at 78 sites all over Austria.

Primary Endpoint:

1. Proof of the effect of 2 years versus 5 years of Anastrozol after 5 years of adjuvant endocrine therapy on the disease free survival

Secondary endpoint:

1. Proof of the effect of 2 years versus 5 years of Anastrozol after 5 years of adjuvant endocrine therapy on the overall survival
2. Comparison of fracture rate in both therapy groups
3. Comparison of incidence of

   1. a secondary carcinoma except the contralateral mammacarcinoma
   2. contralateral mammacarcinoma in both therapie groups

ELIGIBILITY:
Inclusion criteria:

1. Postmenopausal patients with histologically confirmed, local radically treated invasive or minimal-invasiv Mammacarcinom with or without previous chemotherapie and/or radiotherapie.
2. No distant metastasis at randomization
3. No relapse at randomization
4. TNM- classification at time of diagnosis: T1-3, N0 and N+, M0
5. Estrogen- and or progesterone positive before the beginningof primary endocrine therapy
6. Endocrine therapy for 5 years (maximum deviation ±12 months)
7. Therapy break (from the preliminary therapie) maximum 12 months.
8. Informed Consent before the randomisation

Exclusion criteria:

1. Premenopausal patients or patients with non definable menopausal statusat time of randomisation
2. Apparent secondary malignant tumor or status after secondary malignant tumor (Exceptions: simultaniously appearing bilateral breast carcinoma, estrogen- and or progesteronereceptor positive on both sides at the time of diagnosis; in situ carcinomaof the cervix and basal cell carcinoma of the skin)
3. General contraindication respectively hypersensitivity to Anastrozol.
4. In-situ carcinoma of any size with or without Mb. Paget of the Mamilla respectively T4 tumor at the time of first diagnosis.
5. Receptor unknown or negative at time of diagnosis respectively at beginning of primary endocrine therapy
6. Known liver- and/or kidneyinsufficiency
7. Performance Index >2 according to WHO
8. Regular intake of hormon supplement as well as Hormone Replacement Therapy (HRT) more than 6 months since primary surgery of the mamma carcinoma
9. Serious accessory disease, that prevents the adjuvant therapy according to protocol and/or the regular follow-up care.
10. Lacking compliance of the patient
11. Legal incompetence and/or other circumstances, that prevent the patient from understanding the nature, meaning and consequences of the clinical trial
12. Existing psychiatrical diseaseaccording to ICD (especially alcohol addiction) et the time of admission into the study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3484 (Actual)
Dates: Start 2004-03-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Austria Medical Director, MD, Study Director — AstraZeneca
Locations (46):
- Austria (46):
  - Research Site, Amstetten
  - Research Site, Bad Ischl
  - Research Site, Baden
  - Research Site, Bregenz
  - Research Site, Dornbirn
  - Research Site, Eisenstadt
  - Research Site, Feldbach
  - Research Site, Feldkirch
  - Research Site, Freistadt
  - Research Site, Fürstenfeld
  - Research Site, Gmunden
  - Research Site, Graz
  - Research Site, Güssing
  - Research Site, Hainburg an der Donau
  - Research Site, Hall in Tirol
  - Research Site, Innsbruck
  - Research Site, Kirchdorf
  - Research Site, Klagenfurt
  - Research Site, Krems
  - Research Site, Kufstein
  - Research Site, Leoben
  - Research Site, Lienz
  - Research Site, Linz
  - Research Site, Mistelbach
  - Research Site, Mödling
  - Research Site, Neunkirchen
  - Research Site, Oberpullendorf
  - Research Site, Oberwart
  - Research Site, Ried im Innkreis
  - Research Site, Rottenmann
  - Research Site, Salzburg
  - Research Site, Sankt Pölten
  - Research Site, Sankt Veit an der Glan
  - Research Site, Scheibbs
  - Research Site, Schladming
  - Research Site, Schwarzach
  - Research Site, Steyr
  - Research Site, Vienna
  - Research Site, Villach
  - Research Site, Vöcklabruck
  - Research Site, Waidhofen an der Thaya
  - Research Site, Weiz
  - Research Site, Wels
  - Research Site, Wiener Neustadt
  - Research Site, Wolfsberg
  - Research Site, Zams

REFERENCES:
- [Derived] Gnant M, Fitzal F, Rinnerthaler G, Steger GG, Greil-Ressler S, Balic M, Heck D, Jakesz R, Thaler J, Egle D, Manfreda D, Bjelic-Radisic V, Wieder U, Singer CF, Melbinger-Zeinitzer E, Haslbauer F, Sevelda P, Trapl H, Wette V, Wimmer K, Gampenrieder SP, Bartsch R, Kacerovsky-Strobl S, Suppan C, Brunner C, Deutschmann C, Soelkner L, Fesl C, Greil R; Austrian Breast and Colorectal Cancer Study Group. Duration of Adjuvant Aromatase-Inhibitor Therapy in Postmenopausal Breast Cancer. N Engl J Med. 2021 Jul 29;385(5):395-405. doi: 10.1056/NEJMoa2104162. PMID 34320285
- See also: 1033AU/0003 CSP redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2464&filename=1033AU0003_CSP_redacted.pdf
- See also: 1033AU/0003 SAP redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2464&filename=1033AU0003_SAP_redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was randomized Feb 26, 2004, the last patient was randomized June 30, 2010. Randomization took place in 75 Austrian clinical sites. In total, 3,484 patients were enrolled.
Pre-assignment Details: Fourteen patients did not sign the Informed Consent, resulting in 3,470 patients who started the trial.
Period: Overall Study
Arm/Group | Arm A: Anastrozol | Arm B: Anastrozol
Started (ITT: all randomized, signed Informed Consent) | 1732 | 1738
Safety Analysis Set (All randomized, at least one dose) | 1705 | 1710
Completed | 860 | 842
Not Completed | 872 | 896
Not completed — Lost to Follow-up | 9 | 5
Not completed — Withdrawal by Subject | 37 | 50
Not completed — Death | 206 | 207
Not completed — Other reasons | 10 | 9
Not completed — Discontinuation by sponsor | 580 | 593
Not completed — Protocol Violation | 30 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Anastrozol | Arm B: Anastrozol | Total
Number analyzed (Participants) | 1732 | 1738 | 3470
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [58 to 70] | 64 [59 to 69] | 64 [59 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1732 | 1738 | 3470
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
pN-stage [Count of Participants; unit: Participants] — Categories of affected lymph nodes:
  pN0: no affected lymph nodes, pN1: 1-3 affected lymph nodes, pN2: 4-9 affected lymph nodes, pN3: 10 or more affected lymph nodes
  Participants
    pN0 | 1140 | 1162 | 2302
    pN1 | 551 | 523 | 1074
    pN2 | 30 | 41 | 71
    pN3 | 7 | 8 | 15
    Unknown | 4 | 4 | 8
pT-stage [Count of Participants; unit: Participants] — Categories of tumor size:
  pT1: <2 cm, pT2: 2 to 5 cm, pT3: > 5 cm, pTx: not determinable
  Participants
    pT1 | 1254 | 1254 | 2508
    pT2 | 440 | 442 | 882
    pT3 | 30 | 32 | 62
    pTx | 4 | 6 | 10
    Unknown | 4 | 4 | 8
Previous Chemotherapy [Count of Participants; unit: Participants]
  Chemotherapy containing anthracycline | 246 | 236 | 482
  Chemotherapy containing taxane | 93 | 95 | 188
  Other chemotherapy | 167 | 163 | 330
  No chemotherapy | 1224 | 1241 | 2465
  Unknown | 2 | 3 | 5
Previous Endocrine Therapy [Count of Participants; unit: Participants]
  2 years of anti-estrogen + 3 years Anastrozole | 416 | 419 | 835
  5 years of anti-estrogen | 855 | 862 | 1717
  Another, comparable endocrine therapy | 459 | 454 | 913
  Unknown | 2 | 3 | 5
Estrogen Receptor Status [Count of Participants; unit: Participants]
  Negative | 45 | 46 | 91
  Positive (+/++/+++) | 1686 | 1689 | 3375
  Unknown | 1 | 3 | 4
Progesterone Receptor Status [Count of Participants; unit: Participants]
  Negative | 332 | 356 | 688
  Positive (+/++/+++) | 1398 | 1375 | 2773
  Unknown | 2 | 7 | 9
Surgery Type [Count of Participants; unit: Participants]
  Breast-conserving surgery | 1360 | 1405 | 2765
  Modified radical mastectomy | 367 | 319 | 686
  Other | 4 | 12 | 16
  Unknown | 1 | 2 | 3
Sentinel Node Biopsy [Count of Participants; unit: Participants]
  No | 900 | 887 | 1787
  Yes | 820 | 836 | 1656
  Unknown | 12 | 15 | 27
Axillary Surgery [Count of Participants; unit: Participants]
  No | 386 | 405 | 791
  Yes | 1345 | 1331 | 2676
  Unknown | 1 | 2 | 3
Tumor Grading [Count of Participants; unit: Participants] — Grade of differentiation:
  G1: well differentiated (cells look more like normal breast tissue), G2: moderately differentiated, G3: poorly differentiated, GX: not determinable
  Participants
    G1 | 247 | 261 | 508
    G2 | 1107 | 1090 | 2197
    G3 | 326 | 348 | 674
    GX | 27 | 12 | 39
    Unknown | 25 | 27 | 52
Previous Radiotherapy [Count of Participants; unit: Participants]
  No | 356 | 327 | 683
  Yes | 1373 | 1407 | 2780
  Unknown | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival After Prolonged Endocrine Treatment
Description: To determine whether 5 years of additional Anastrozole was more effective than 2 years of additional Anastrozole after 5 years of adjuvant endocrine therapy in terms of disease-free survival.
Time Frame: DFS was defined as the time from two years after randomization to the earliest occurrence of loco-regional recurrence, distant recurrence, contralateral new breast cancer, second cancer or death from any cause, assessed up to a maximum of 8.5 years
Population: Per-Protocol (PP) Population, defined as all randomized patients who signed the informed consent who complied with the inclusion and exclusion criteria, who had at least one follow-up examination after randomization and who survived without recurrence for two years.
Measure: Median (Inter-Quartile Range); unit: Years
Arm/Group | Arm A: Anastrozol | Arm B: Anastrozol
Number analyzed (Participants) | 1281 | 1323
Years | NA [7.7 to NA] — NA - Not applicable, estimates cannot be calculated due to too few events. | NA [8.1 to NA] — NA - Not applicable, estimates cannot be calculated due to too few events.
Statistical Analysis 1: Comparison: Arm A: Anastrozol vs Arm B: Anastrozol; Arm A: Anastrozole for 2 yerars Arm B: Anastrozole for 5 years Null hypothesis: there is no difference between the two treatment arms in the probability of a DFS event; Test type: Superiority; p = 0.425, Log Rank; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.79 to 1.11]

2. Secondary Outcome: Overall Survival After Prolonged Endocrine Treatment
Description: To determine whether 5 years of additional Anastrozole was more effective than 2 years of additional Anastrozole after 5 years of adjuvant endocrine therapy in terms of overall survival.
Time Frame: Overall survival was defined as the time from two years after randomization to death due to any cause, assessed up to a maximum of 8.5 years
Population: All randomized patients who signed the informed consent and who did not die during two first two years
Measure: Median (Inter-Quartile Range); unit: Years
Arm/Group | Arm A: Anastrozol | Arm B: Anastrozol
Number analyzed (Participants) | 1665 | 1670
Years | NA [NA to NA] — NA - Not applicable, estimates cannot be calculated due to too few events. | NA [NA to NA] — NA - Not applicable, estimates cannot be calculated due to too few events.
Statistical Analysis 1: Comparison: Arm A: Anastrozol vs Arm B: Anastrozol; Arm A: Anastrozole for 2 yerars Arm B: Anastrozole for 5 years Null hypothesis: there is no difference between the two treatment arms in the probability of a death event; Test type: Superiority; p = 0.867, Log Rank; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.83 to 1.25]

3. Secondary Outcome: Time to First Clinical Fracture
Description: To determine the effect of 2 years versus 5 years of additional Anastrozole after 5 years of adjuvant endocrine therapy on the time to first clinical fracture. Patients without clinical fractures where censored at their last therapy visit (approximately 5 years after randomization).
Time Frame: Time to first clinical fracture was defined as time to first clinical fracture, in the period from 2 years until 5 years after randomization for each patient.
Population: All randomized patients who signed the informed consent and who had no fractures during the first two years
Measure: Median (Inter-Quartile Range); unit: Years
Arm/Group | Arm A: Anastrozol | Arm B: Anastrozol
Number analyzed (Participants) | 1555 | 1570
Years | NA [NA to NA] — NA - Not applicable, estimates cannot be calculated due to too few events. | NA [NA to NA] — NA - Not applicable, estimates cannot be calculated due to too few events.
Statistical Analysis 1: Comparison: Arm A: Anastrozol vs Arm B: Anastrozol; Arm A: Anastrozole for 2 yerars Arm B: Anastrozole for 5 years Null hypothesis: there is no difference between the two treatment arms in the probability of a fracture; Test type: Superiority; p = 0.052, Log Rank; Hazard Ratio (HR) = 1.35, 95% CI 2-sided [1.00 to 1.84]

4. Secondary Outcome: Time to Secondary Carcinoma
Description: To determine whether 5 years of additional Anastrozole was more effective than 2 years of additional Anastrozole after 5 years of adjuvant endocrine therapy in terms of lowering the risk of secondary carcinoma. Subjects without secondary cancer event were censored at the last date when they were known to be secondary cancer free.
Time Frame: Risk of secondary carcinoma was defined as the time from two years after randomization to first occurrence of new secondary cancer without new breast cancer (local or contralateral), assessed up to a maximum of 8.5 years
Population: All randomized patients who signed the informed consent and had no secondary carcinoma (excluding contralateral mammacarcinoma) during the first two years
Measure: Median (Inter-Quartile Range); unit: Years
Arm/Group | Arm A: Anastrozol | Arm B: Anastrozol
Number analyzed (Participants) | 1620 | 1620
Years | NA [NA to NA] — NA - Not applicable, estimates cannot be calculated due to too few events. | NA [NA to NA] — NA - Not applicable, estimates cannot be calculated due to too few events.
Statistical Analysis 1: Comparison: Arm A: Anastrozol vs Arm B: Anastrozol; Arm A: Anastrozole for 2 yerars Arm B: Anastrozole for 5 years Null hypothesis: there is no difference between the two treatment arms in the probability of the occurrence of secondary carcinoma; Test type: Superiority; p = 0.678, Log Rank; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.81 to 1.38]

5. Secondary Outcome: Time to Contralateral Breast Cancer
Description: To determine whether 5 years of additional Anastrozole was more effective than 2 years of additional Anastrozole after 5 years of adjuvant endocrine therapy in terms of lowering the risk of contralateral breast cancer. Subjects without contralateral breast cancer event were censored at the last date when they were known to be contralateral breast cancer free.
Time Frame: Risk of contralateral breast cancer was defined as the time from two years after randomization to first occurrence of new contralateral breast cancer, assessed up to a maximum of 8.5 years
Population: All randomized patients who signed the informed consent and had no contralateral mammacarcinoma during the first two years
Measure: Median (Inter-Quartile Range); unit: Years
Arm/Group | Arm A: Anastrozol | Arm B: Anastrozol
Number analyzed (Participants) | 1636 | 1641
Years | NA [NA to NA] — NA - Not applicable, estimates cannot be calculated due to too few events. | NA [NA to NA] — NA - Not applicable, estimates cannot be calculated due to too few events.
Statistical Analysis 1: Comparison: Arm A: Anastrozol vs Arm B: Anastrozol; Arm A: Anastrozole for 2 years Arm B: Anastrozole for 5 years Null hypothesis: there is no difference between the two treatment arms in the probability of the occurrence of contralateral mammacarcinoma; Test type: Superiority; p = 0.531, Log Rank; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.75 to 1.77]

ADVERSE EVENTS:
Time Frame: Maximum observation period per patient 10.5 years; reporting period for all-cause mortality starts with randomization; adverse event reporting starts with first dose of treatment
Description: All-cause mortality data presented for intention-to-treat analysis set and for the entire study. Serious adverse events (SAEs) reported during treatment phase plus 30 days, and after this period only if the investigator could not preclude a causal link to treatment with Anastrozole. SAEs are based on the safety population (randomized and received at least one dose of study treatment). Other adverse events were not collected in the safety database and are therefore not reported here.
Groups:
- Arm B: Anastrozol - 1 mg Per Day for 5 Years; Arm A: Anastrozol - 1 mg Per Day for 2 Years: Description (Arm-group)
Arm/Group | Arm B: Anastrozol - 1 mg Per Day for 5 Years | Arm A: Anastrozol - 1 mg Per Day for 2 Years
All-Cause Mortality (participants affected / at risk) | 207/1738 | 207/1732
Serious Adverse Events (participants affected / at risk) | 687/1710 | 452/1705
Other Adverse Events (participants affected / at risk) | 0/1710 | 0/1705
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm B: Anastrozol - 1 mg Per Day for 5 Years (N=1710) | Arm A: Anastrozol - 1 mg Per Day for 2 Years (N=1705)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 1 (2)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Bone marrow oedema (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Lymph node calcification (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 (6) | 0 (0)
Mastocytosis (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (2) | 1 (2)
Angina pectoris (Cardiac disorders) | 4 (6) | 4 (9)
Aortic valve disease (Cardiac disorders) | 0 (0) | 1 (2)
Aortic valve prolapse (Cardiac disorders) | 1 (2) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 2 (3) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (2) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 17 (37) | 6 (10)
Atrial flutter (Cardiac disorders) | 1 (2) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (2) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 2 (4) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (2) | 2 (4)
Cardiac arrest (Cardiac disorders) | 1 (3) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (3)
Cardiac failure (Cardiac disorders) | 7 (15) | 6 (12)
Cardiac flutter (Cardiac disorders) | 1 (2) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (2) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (2) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (2)
Cor pulmonale chronic (Cardiac disorders) | 1 (4) | 0 (0)
Coronary artery disease (Cardiac disorders) | 8 (17) | 6 (13)
Intracardiac thrombus (Cardiac disorders) | 1 (2) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 2 (4) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (2)
Mitral valve disease mixed (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 4 (7) | 0 (0)
Myocardial infarction (Cardiac disorders) | 4 (8) | 2 (3)
Myocardial ischaemia (Cardiac disorders) | 1 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 2 (4) | 1 (2)
Sinus node dysfunction (Cardiac disorders) | 1 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (2) | 1 (2)
Tachycardia (Cardiac disorders) | 1 (1) | 3 (9)
Tachycardia paroxysmal (Cardiac disorders) | 0 (0) | 1 (2)
Tricuspid valve incompetence (Cardiac disorders) | 1 (2) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (2) | 1 (2)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (3)
Wolff-parkinson-white syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 0 (0) | 1 (2)
Anomalous arrangement of pancreaticobiliary duct (Congenital, familial and genetic disorders) | 1 (2) | 0 (0)
Choledochal cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (2)
Congenital uterine anomaly (Congenital, familial and genetic disorders) | 1 (2) | 0 (0)
Corneal opacity congenital (Congenital, familial and genetic disorders) | 1 (2) | 0 (0)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Epidermal naevus (Congenital, familial and genetic disorders) | 0 (0) | 1 (2)
Foramen magnum stenosis (Congenital, familial and genetic disorders) | 1 (2) | 0 (0)
Cupulolithiasis (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Deafness (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 2 (4)
Inner ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (2) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 2 (3) | 2 (4)
Tympanosclerosis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 8 (15) | 5 (9)
Vertigo positional (Ear and labyrinth disorders) | 2 (3) | 2 (4)
Goitre (Endocrine disorders) | 12 (22) | 4 (8)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (2)
Hyperparathyroidism primary (Endocrine disorders) | 2 (3) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 3 (6) | 1 (2)
Thyroid haemorrhage (Endocrine disorders) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 2 (3)
Age-related macular degeneration (Eye disorders) | 1 (2) | 0 (0)
Astigmatism (Eye disorders) | 1 (3) | 0 (0)
Blepharochalasis (Eye disorders) | 2 (4) | 0 (0)
Cataract (Eye disorders) | 26 (68) | 12 (26)
Cataract cortical (Eye disorders) | 4 (10) | 0 (0)
Cataract nuclear (Eye disorders) | 2 (5) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 1 (2)
Exfoliation syndrome (Eye disorders) | 0 (0) | 1 (2)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (2) | 1 (2)
Lens dislocation (Eye disorders) | 1 (1) | 0 (0)
Macular degeneration (Eye disorders) | 1 (2) | 2 (4)
Macular hole (Eye disorders) | 3 (6) | 0 (0)
Maculopathy (Eye disorders) | 1 (1) | 1 (2)
Myopia (Eye disorders) | 1 (3) | 0 (0)
Photopsia (Eye disorders) | 1 (2) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (3)
Retinal degeneration (Eye disorders) | 1 (2) | 0 (0)
Retinal detachment (Eye disorders) | 2 (4) | 0 (0)
Retinal disorder (Eye disorders) | 1 (2) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (2)
Retinal tear (Eye disorders) | 1 (2) | 0 (0)
Retinopathy hypertensive (Eye disorders) | 1 (2) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (2) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 13 (22) | 4 (12)
Abdominal pain lower (Gastrointestinal disorders) | 1 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (7) | 2 (5)
Abdominal symptom (Gastrointestinal disorders) | 1 (2) | 0 (0)
Abdominal wall disorder (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abnormal faeces (Gastrointestinal disorders) | 1 (2) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 1 (2) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 1 (2) | 1 (2)
Anal polyp (Gastrointestinal disorders) | 1 (2) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 1 (2) | 0 (0)
Anorectal disorder (Gastrointestinal disorders) | 1 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (2) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Coeliac disease (Gastrointestinal disorders) | 1 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (2)
Colitis microscopic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 2 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (7) | 2 (2)
Dental alveolar anomaly (Gastrointestinal disorders) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 12 (21) | 6 (11)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (2) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 1 (2)
Diverticulum intestinal (Gastrointestinal disorders) | 6 (12) | 2 (3)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Enterocele (Gastrointestinal disorders) | 0 (0) | 2 (4)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastric polyps (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (4)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (5) | 5 (10)
Gastritis erosive (Gastrointestinal disorders) | 1 (2) | 1 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (4) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (10) | 3 (6)
Haematochezia (Gastrointestinal disorders) | 2 (3) | 4 (7)
Haemorrhoids (Gastrointestinal disorders) | 5 (10) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 3 (5) | 2 (4)
Ileus (Gastrointestinal disorders) | 2 (4) | 1 (1)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (4) | 2 (4)
Intestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (2)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (2)
Intestinal prolapse (Gastrointestinal disorders) | 1 (2) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (2) | 1 (2)
Large intestine polyp (Gastrointestinal disorders) | 16 (28) | 8 (17)
Mallory-weiss syndrome (Gastrointestinal disorders) | 1 (2) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (2)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (13) | 4 (14)
Oesophagitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (4) | 1 (2)
Pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 1 (2)
Proctitis (Gastrointestinal disorders) | 2 (6) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 5 (10) | 1 (2)
Subileus (Gastrointestinal disorders) | 1 (2) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 1 (4)
Umbilical hernia (Gastrointestinal disorders) | 1 (2) | 2 (3)
Vomiting (Gastrointestinal disorders) | 4 (8) | 3 (10)
Asthenia (General disorders) | 1 (2) | 0 (0)
Calcinosis (General disorders) | 1 (2) | 1 (2)
Chest discomfort (General disorders) | 0 (0) | 2 (3)
Chest pain (General disorders) | 9 (19) | 4 (6)
Condition aggravated (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 6 (12) | 0 (0)
Fat necrosis (General disorders) | 1 (2) | 1 (2)
Fatigue (General disorders) | 1 (2) | 1 (2)
Fibrosis (General disorders) | 0 (0) | 1 (2)
General physical health deterioration (General disorders) | 1 (4) | 4 (7)
Hernia (General disorders) | 1 (2) | 0 (0)
Hyperplasia (General disorders) | 0 (0) | 2 (4)
Ill-defined disorder (General disorders) | 1 (2) | 0 (0)
Impaired healing (General disorders) | 4 (8) | 1 (2)
Implant site extravasation (General disorders) | 0 (0) | 1 (1)
Implant site fibrosis (General disorders) | 1 (2) | 0 (0)
Incarcerated hernia (General disorders) | 0 (0) | 1 (2)
Inflammation (General disorders) | 0 (0) | 1 (2)
Multiple organ dysfunction syndrome (General disorders) | 1 (2) | 0 (0)
Oedema mucosal (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (2) | 0 (0)
Peripheral swelling (General disorders) | 1 (2) | 0 (0)
Polyp (General disorders) | 1 (2) | 1 (2)
Pyrexia (General disorders) | 4 (8) | 2 (4)
Sudden cardiac death (General disorders) | 1 (2) | 0 (0)
Ampulla of vater stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 2 (4) | 1 (2)
Biliary tract disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 3 (6) | 2 (4)
Cholecystitis acute (Hepatobiliary disorders) | 1 (2) | 2 (3)
Cholecystitis chronic (Hepatobiliary disorders) | 4 (5) | 1 (2)
Cholelithiasis (Hepatobiliary disorders) | 14 (27) | 15 (27)
Gallbladder disorder (Hepatobiliary disorders) | 1 (2) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 1 (2) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (2) | 1 (2)
Hepatitis cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (2)
Jaundice (Hepatobiliary disorders) | 1 (4) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (2)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (2)
Abscess of salivary gland (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (2) | 0 (0)
Appendicitis (Infections and infestations) | 2 (4) | 1 (2)
Bronchitis (Infections and infestations) | 3 (5) | 3 (4)
Campylobacter gastroenteritis (Infections and infestations) | 1 (2) | 0 (0)
Chest wall abscess (Infections and infestations) | 1 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (2)
Diverticulitis (Infections and infestations) | 5 (13) | 7 (16)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 (0) | 1 (2)
Ear infection (Infections and infestations) | 1 (2) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 1 (2)
Erysipelas (Infections and infestations) | 6 (13) | 7 (10)
Extradural abscess (Infections and infestations) | 1 (2) | 0 (0)
Fungal infection (Infections and infestations) | 1 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (7) | 3 (6)
Helicobacter gastritis (Infections and infestations) | 3 (3) | 1 (2)
Herpes zoster (Infections and infestations) | 1 (2) | 0 (0)
Infected dermal cyst (Infections and infestations) | 1 (2) | 0 (0)
Intervertebral discitis (Infections and infestations) | 1 (2) | 0 (0)
Meningitis viral (Infections and infestations) | 1 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (2)
Neuroborreliosis (Infections and infestations) | 1 (2) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 1 (2) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 2 (3)
Pharyngitis (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 11 (22) | 5 (12)
Pyelonephritis (Infections and infestations) | 1 (1) | 2 (4)
Pyometra (Infections and infestations) | 0 (0) | 1 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (5)
Rhinitis (Infections and infestations) | 1 (2) | 0 (0)
Salpingitis (Infections and infestations) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (2)
Sinobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 2 (4)
Skin infection (Infections and infestations) | 1 (2) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (2) | 0 (0)
Urethral carbuncle (Infections and infestations) | 1 (2) | 1 (2)
Urinary tract infection (Infections and infestations) | 11 (23) | 0 (0)
Urosepsis (Infections and infestations) | 1 (2) | 1 (2)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (2)
Vestibular neuronitis (Infections and infestations) | 2 (2) | 0 (0)
Vulval abscess (Infections and infestations) | 0 (0) | 1 (2)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 20 (38) | 5 (9)
Bankart lesion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 1 (2) | 1 (2)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (4)
Concussion (Injury, poisoning and procedural complications) | 2 (4) | 3 (6)
Contusion (Injury, poisoning and procedural complications) | 10 (18) | 4 (10)
Coronary bypass thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Facial bones fracture (Injury, poisoning and procedural complications) | 2 (4) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 2 (4)
Femoral neck fracture (Injury, poisoning and procedural complications) | 5 (9) | 2 (4)
Femur fracture (Injury, poisoning and procedural complications) | 8 (12) | 3 (6)
Fibula fracture (Injury, poisoning and procedural complications) | 2 (4) | 1 (2)
Foot fracture (Injury, poisoning and procedural complications) | 4 (8) | 7 (14)
Forearm fracture (Injury, poisoning and procedural complications) | 2 (4) | 3 (5)
Fracture (Injury, poisoning and procedural complications) | 3 (5) | 3 (4)
Fractured sacrum (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 6 (12) | 2 (4)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Hip fracture (Injury, poisoning and procedural complications) | 3 (5) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 13 (24) | 5 (8)
Ilium fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 6 (10) | 2 (4)
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (6) | 1 (1)
Keratorhexis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3 (6) | 5 (11)
Meniscus injury (Injury, poisoning and procedural complications) | 14 (27) | 4 (8)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Overdose (Injury, poisoning and procedural complications) | 1 (4) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (2) | 1 (2)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Postoperative wound complication (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 4 (7) | 1 (4)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 29 (55) | 21 (40)
Rib fracture (Injury, poisoning and procedural complications) | 3 (4) | 4 (6)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (2) | 2 (3)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 3 (6) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (4)
Suture related complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (4)
Tendon rupture (Injury, poisoning and procedural complications) | 4 (6) | 2 (4)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 3 (6) | 3 (5)
Tibia fracture (Injury, poisoning and procedural complications) | 5 (8) | 3 (4)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (4) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 2 (2) | 1 (2)
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 3 (5) | 1 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 5 (8) | 4 (7)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 4 (7) | 1 (2)
Angiogram (Investigations) | 1 (2) | 0 (0)
Biopsy lymph gland (Investigations) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 2 (3) | 0 (0)
Blood glucose abnormal (Investigations) | 1 (2) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (2)
Bronchoscopy (Investigations) | 0 (0) | 1 (1)
Carcinoembryonic antigen increased (Investigations) | 1 (2) | 0 (0)
Colonoscopy (Investigations) | 1 (1) | 0 (0)
Electrocardiogram change (Investigations) | 0 (0) | 1 (2)
Endoscopic retrograde cholangiopancreatography (Investigations) | 0 (0) | 1 (2)
Endoscopy upper gastrointestinal tract (Investigations) | 1 (1) | 0 (0)
Lipids abnormal (Investigations) | 1 (2) | 0 (0)
Liver function test increased (Investigations) | 1 (2) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (2) | 0 (0)
Smear cervix abnormal (Investigations) | 1 (4) | 1 (4)
Tumour marker increased (Investigations) | 1 (2) | 0 (0)
Varicella virus test positive (Investigations) | 1 (2) | 0 (0)
Weight decreased (Investigations) | 1 (2) | 1 (2)
Calciphylaxis (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 1 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (6) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Obesity (Metabolism and nutrition disorders) | 1 (2) | 2 (4)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (10) | 2 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (13) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (6)
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2)
Foot deformity (Musculoskeletal and connective tissue disorders) | 14 (28) | 14 (30)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 15 (29) | 9 (15)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (4)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (6) | 3 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (3)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Myosclerosis (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 74 (164) | 29 (60)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 4 (8) | 3 (8)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (7) | 3 (7)
Plica syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (2) | 5 (9)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Spinal fusion acquired (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (6)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 5 (10) | 2 (2)
Synovitis (Musculoskeletal and connective tissue disorders) | 3 (6) | 1 (2)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (6)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (2)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (6) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 2 (4)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 2 (3)
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (19) | 2 (4)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (6) | 0 (0)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (4)
Breast angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (22) | 2 (3)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 0 (0)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Carcinoid tumour of the caecum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid tumour of the stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Cardiac neoplasm unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (2)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 3 (5)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (8) | 4 (7)
Diffuse large b-cell lymphoma stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Enchondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (6) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Fallopian tube cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Glomus tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Haemangioma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Intra-abdominal haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (2)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (2)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (6)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (12) | 3 (4)
Malignant melanoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Malignant neoplasm of uterine adnexa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3)
Meningeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 1 (2)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Metastases to breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Mucinous breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 1 (2)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (2)
Oral fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 0 (0)
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 3 (5)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rosai-dorfman syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Sarcoma uterus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 0 (0)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (6) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (4)
Superficial spreading melanoma stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 0 (0)
Tongue neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (15) | 1 (1)
Ataxia (Nervous system disorders) | 1 (2) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 1 (2) | 0 (0)
Burning feet syndrome (Nervous system disorders) | 1 (2) | 0 (0)
Carotid artery aneurysm (Nervous system disorders) | 0 (0) | 1 (2)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (2)
Carpal tunnel syndrome (Nervous system disorders) | 10 (18) | 10 (23)
Cerebral haemorrhage (Nervous system disorders) | 2 (4) | 0 (0)
Cerebral infarction (Nervous system disorders) | 3 (5) | 2 (5)
Cerebral ischaemia (Nervous system disorders) | 2 (3) | 1 (2)
Cerebrovascular accident (Nervous system disorders) | 5 (12) | 1 (2)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 4 (8) | 1 (2)
Dementia (Nervous system disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 2 (7)
Dysaesthesia (Nervous system disorders) | 1 (2) | 0 (0)
Embolic cerebral infarction (Nervous system disorders) | 1 (2) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (2) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (2)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (2)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (4) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (2) | 1 (4)
Horner's syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Hypertonia (Nervous system disorders) | 1 (2) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (2)
Intracranial aneurysm (Nervous system disorders) | 1 (2) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (2)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (4)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Mental impairment (Nervous system disorders) | 1 (2) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (2) | 0 (0)
Nerve root compression (Nervous system disorders) | 0 (0) | 1 (2)
Neuromuscular blockade (Nervous system disorders) | 1 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (4) | 0 (0)
Paralysis (Nervous system disorders) | 1 (2) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 2 (4)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 1 (2) | 3 (4)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (2)
Quadriparesis (Nervous system disorders) | 0 (0) | 1 (2)
Radicular pain (Nervous system disorders) | 1 (1) | 1 (2)
Ruptured cerebral aneurysm (Nervous system disorders) | 0 (0) | 1 (2)
Sciatica (Nervous system disorders) | 10 (20) | 9 (17)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 9 (17) | 3 (5)
Tension headache (Nervous system disorders) | 0 (0) | 1 (2)
Thalamic infarction (Nervous system disorders) | 2 (4) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 8 (15) | 2 (2)
Trigeminal neuralgia (Nervous system disorders) | 1 (2) | 0 (0)
Vertigo cns origin (Nervous system disorders) | 1 (2) | 0 (0)
Visual pathway disorder (Nervous system disorders) | 0 (0) | 1 (1)
Vocal cord paresis (Nervous system disorders) | 1 (2) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 1 (1)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 2 (6)
Anxiety disorder (Psychiatric disorders) | 1 (2) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (2) | 1 (2)
Burnout syndrome (Psychiatric disorders) | 0 (0) | 1 (2)
Completed suicide (Psychiatric disorders) | 0 (0) | 2 (3)
Depression (Psychiatric disorders) | 7 (13) | 6 (12)
Insomnia (Psychiatric disorders) | 1 (2) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 1 (2)
Major depression (Psychiatric disorders) | 1 (4) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (2) | 1 (2)
Persistent depressive disorder (Psychiatric disorders) | 2 (3) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 0 (0) | 1 (2)
Schizoaffective disorder depressive type (Psychiatric disorders) | 0 (0) | 1 (6)
Somatic symptom disorder (Psychiatric disorders) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 1 (2)
Haematuria (Renal and urinary disorders) | 3 (5) | 2 (4)
Hydronephrosis (Renal and urinary disorders) | 2 (4) | 0 (0)
Micturition disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (3) | 3 (6)
Renal aneurysm (Renal and urinary disorders) | 1 (2) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 1 (2) | 0 (0)
Renal colic (Renal and urinary disorders) | 2 (3) | 1 (2)
Renal cyst (Renal and urinary disorders) | 2 (4) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (6) | 2 (4)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 2 (4) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 1 (2) | 0 (0)
Urethral haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 4 (8) | 1 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (2)
Adenomyosis (Reproductive system and breast disorders) | 1 (2) | 1 (6)
Adnexa uteri cyst (Reproductive system and breast disorders) | 2 (5) | 2 (3)
Breast calcifications (Reproductive system and breast disorders) | 5 (10) | 4 (6)
Breast disorder (Reproductive system and breast disorders) | 2 (4) | 0 (0)
Breast fibrosis (Reproductive system and breast disorders) | 1 (2) | 1 (2)
Breast hyperplasia (Reproductive system and breast disorders) | 1 (2) | 1 (2)
Breast mass (Reproductive system and breast disorders) | 2 (3) | 1 (1)
Breast necrosis (Reproductive system and breast disorders) | 1 (1) | 1 (2)
Cervical dysplasia (Reproductive system and breast disorders) | 2 (4) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Colpocele (Reproductive system and breast disorders) | 0 (0) | 2 (3)
Cystocele (Reproductive system and breast disorders) | 3 (6) | 2 (4)
Ectropion of cervix (Reproductive system and breast disorders) | 0 (0) | 1 (4)
Endometrial atrophy (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Endometrial disorder (Reproductive system and breast disorders) | 4 (12) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 16 (39) | 6 (16)
Endometrial metaplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hydrometra (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (3)
Menorrhagia (Reproductive system and breast disorders) | 1 (2) | 1 (2)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (6)
Nipple exudate bloody (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Ovarian cyst (Reproductive system and breast disorders) | 8 (17) | 4 (17)
Ovarian disorder (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 11 (22) | 9 (19)
Rectocele (Reproductive system and breast disorders) | 1 (2) | 3 (6)
Uterine disorder (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 16 (51) | 6 (17)
Uterine prolapse (Reproductive system and breast disorders) | 2 (4) | 2 (4)
Uterovaginal prolapse (Reproductive system and breast disorders) | 5 (10) | 2 (3)
Vaginal cyst (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Vaginal dysplasia (Reproductive system and breast disorders) | 1 (4) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (2) | 7 (12)
Vaginal polyp (Reproductive system and breast disorders) | 2 (3) | 1 (4)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (2) | 2 (4)
Vaginal stricture (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulva cyst (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial polyp (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (11) | 3 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (17) | 3 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (2)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Nasal turbinate abnormality (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 1 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 14 (27) | 4 (8)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary vascular disorder (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (7) | 2 (4)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (12)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (6)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Sebaceous gland disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 (7) | 1 (2)
Urticaria chronic (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Alcohol rehabilitation (Surgical and medical procedures) | 1 (2) | 0 (0)
Angioplasty (Surgical and medical procedures) | 1 (2) | 0 (0)
Aortic valve replacement (Surgical and medical procedures) | 1 (3) | 0 (0)
Arthrodesis (Surgical and medical procedures) | 0 (0) | 1 (1)
Breast operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Breast reconstruction (Surgical and medical procedures) | 0 (0) | 1 (1)
Bunion operation (Surgical and medical procedures) | 2 (3) | 0 (0)
Cancer surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 (2) | 0 (0)
Carpal tunnel decompression (Surgical and medical procedures) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 2 (6) | 3 (5)
Central venous catheter removal (Surgical and medical procedures) | 2 (3) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Colostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Enterostomy (Surgical and medical procedures) | 0 (0) | 1 (2)
Eye operation (Surgical and medical procedures) | 1 (2) | 0 (0)
Gastric banding (Surgical and medical procedures) | 1 (2) | 0 (0)
Hernia repair (Surgical and medical procedures) | 1 (2) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 1 (2) | 4 (6)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Hysterosalpingo-oophorectomy (Surgical and medical procedures) | 0 (0) | 1 (2)
Intraocular lens implant (Surgical and medical procedures) | 2 (6) | 0 (0)
Jaw operation (Surgical and medical procedures) | 1 (2) | 0 (0)
Joint arthroplasty (Surgical and medical procedures) | 2 (2) | 1 (2)
Knee arthroplasty (Surgical and medical procedures) | 5 (10) | 3 (6)
Knee operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Large intestinal polypectomy (Surgical and medical procedures) | 1 (2) | 0 (0)
Lipoma excision (Surgical and medical procedures) | 2 (4) | 1 (2)
Lithotripsy (Surgical and medical procedures) | 0 (0) | 1 (2)
Lymphadenectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Mammoplasty (Surgical and medical procedures) | 1 (2) | 2 (4)
Medical device removal (Surgical and medical procedures) | 0 (0) | 1 (2)
Mole excision (Surgical and medical procedures) | 1 (2) | 0 (0)
Nasal operation (Surgical and medical procedures) | 1 (2) | 0 (0)
Nephrectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Oophorectomy (Surgical and medical procedures) | 0 (0) | 1 (2)
Oophorectomy bilateral (Surgical and medical procedures) | 1 (2) | 0 (0)
Plastic surgery (Surgical and medical procedures) | 1 (2) | 0 (0)
Posterior lens capsulotomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Postoperative care (Surgical and medical procedures) | 0 (0) | 1 (2)
Radioactive iodine therapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Rectal polypectomy (Surgical and medical procedures) | 1 (2) | 0 (0)
Renal cyst excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Salpingo-oophorectomy bilateral (Surgical and medical procedures) | 1 (2) | 0 (0)
Scar excision (Surgical and medical procedures) | 2 (4) | 0 (0)
Skin graft (Surgical and medical procedures) | 1 (2) | 0 (0)
Spinal decompression (Surgical and medical procedures) | 0 (0) | 1 (2)
Spinal operation (Surgical and medical procedures) | 1 (2) | 0 (0)
Synovectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Synovial cyst removal (Surgical and medical procedures) | 0 (0) | 1 (2)
Tendon operation (Surgical and medical procedures) | 1 (2) | 0 (0)
Thyreostatic therapy (Surgical and medical procedures) | 1 (2) | 0 (0)
Thyroidectomy (Surgical and medical procedures) | 2 (3) | 0 (0)
Toe operation (Surgical and medical procedures) | 2 (4) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Uterine tumour excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Vaginoperineoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Varicose vein operation (Surgical and medical procedures) | 0 (0) | 1 (2)
Aortic aneurysm (Vascular disorders) | 2 (4) | 1 (2)
Aortic arteriosclerosis (Vascular disorders) | 1 (2) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (2) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (2) | 1 (2)
Blood pressure fluctuation (Vascular disorders) | 1 (2) | 0 (0)
Blood pressure inadequately controlled (Vascular disorders) | 1 (2) | 0 (0)
Circulatory collapse (Vascular disorders) | 2 (4) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 7 (15) | 3 (5)
Embolism (Vascular disorders) | 0 (0) | 1 (2)
Embolism arterial (Vascular disorders) | 1 (4) | 1 (2)
Extrinsic iliac vein compression (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 2 (4) | 2 (4)
Hypertension (Vascular disorders) | 8 (14) | 6 (10)
Hypertensive crisis (Vascular disorders) | 13 (27) | 1 (2)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (2)
Intermittent claudication (Vascular disorders) | 1 (4) | 0 (0)
Lymphoedema (Vascular disorders) | 3 (8) | 2 (3)
Orthostatic hypotension (Vascular disorders) | 2 (3) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (4) | 1 (2)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (2)
Peripheral artery stenosis (Vascular disorders) | 2 (4) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 4 (8)
Subclavian artery stenosis (Vascular disorders) | 1 (2) | 0 (0)
Temporal arteritis (Vascular disorders) | 0 (0) | 1 (2)
Thrombosis (Vascular disorders) | 3 (8) | 1 (1)
Varicose vein (Vascular disorders) | 8 (15) | 12 (27)
Vasculitis (Vascular disorders) | 0 (0) | 1 (3)
Vein disorder (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 4 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI/Sponsor collaborate in good faith regarding contents/formation of any PI publication/disclosure; PI pays due consideration to comments/opinions of Sponsor. Prior to any publication PI undertakes to provide Sponsor with preliminary data and drafts of publication/disclosures (oral or written) and with proposed final manuscript. Sponsor can review within 30 days and can require that submission for publication/disclosure of manuscript be delayed in order for Sponsor to file patent applications.

DOCUMENTS (2):
  • Study Protocol (2009-11-27): https://cdn.clinicaltrials.gov/large-docs/20/NCT00295620/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT00295620/SAP_001.pdf